CLINICAL TRIAL: NCT07044674
Title: Cataract Surgery: Randomized Comparative Clinical Trial
Brief Title: A Cataract Surgery Clinical Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor's business decision based on strategic shifts
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTV678-P002
Record Dates: First submitted 2025-06-24; First posted 2025-07-01 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Cataract
Keywords: Phacoemulsification; Anterior segment
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- UNITY Vitreoretinal Cataract System (VCS) (Experimental): Anterior segment ophthalmic surgery in one eye using UNITY Vitreoretinal Cataract System (VCS)
  Interventions: Device: UNITY Vitreoretinal Cataract System; Procedure: Anterior segment ophthalmic surgery
- CENTURION Vision System with Active Sentry (CAS) (Active Comparator): Anterior segment ophthalmic surgery in one eye using CENTURION Vision System with Active Sentry (CAS)
  Interventions: Device: CENTURION Vision System with Active Sentry; Procedure: Anterior segment ophthalmic surgery

INTERVENTIONS:
Device: UNITY Vitreoretinal Cataract System — UNITY VCS is a commercially approved surgical system that facilitates the management of fluid and gases, as well as removal, grasping, cutting, illumination, and coagulation of ocular materials during eye surgery. It consists of a console, remote control, foot controller, video overlay, and compatible anterior segment devices. In this study, it will be used for the removal of cataracts.
  Other Names: VCS
  Arms: UNITY Vitreoretinal Cataract System (VCS)
Device: CENTURION Vision System with Active Sentry — CAS is a commercially approved surgical system for use during anterior segment ophthalmic surgery. It consists of a console, foot controller, remote control, video overlay, and compatible anterior segment devices. The Active Sentry handpiece will be used.
  Other Names: CAS
  Arms: CENTURION Vision System with Active Sentry (CAS)
Procedure: Anterior segment ophthalmic surgery — Cataract surgery during which the crystalline lens (often cloudy) is broken into small pieces and gently removed from the eye with suction (phacoemulsification)

SUMMARY:
The purpose of the study is to compare the efficiency and safety of UNITY™ Vitreoretinal Cataract System (UNITY VCS) to CENTURION® Vision System with Active Sentry (CAS) in adult subjects with grade 2 or greater nuclear sclerotic cataracts who require phacoemulsification in both eyes. Subjects will attend a total of 8 scheduled visits for an individual duration of participation of approximately 1 month.

DETAILED DESCRIPTION:
In this contralateral eye clinical study, one eye will undergo surgery with UNITY VCS and the other eye will undergo surgery with CAS. The second eye surgery will occur 0 to 14 days after the first eye surgery.

ELIGIBILITY:
Key Inclusion Criteria:

* Clinically documented diagnosis of age-related nuclear sclerotic cataract of grade 2 or greater in both eyes;
* Both eyes with similar nuclear sclerotic cataract severity and type (within 1 cataract grade);
* Both eyes able to be implanted with same intraocular lens material;
* Both eyes able to receive the same ophthalmic viscosurgical device (OVD).
* Other protocol-specified inclusion criteria may apply.

Key Exclusion Criteria:

* Planned intraoperative glaucoma surgery or expected postoperative procedures during the study in either study eye;
* Laser-assisted cataract surgery in either study eye;
* Any ocular disease and/or condition that, in the investigator's clinical judgement, may put the subject at significant risk, may compromise study results, or may interfere significantly with the subject's participation in the study.
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Cumulative Dissipated Energy (CDE) | Day 0 surgery, each eye
  Cumulative Dissipated Energy (CDE) is the measure of energy released at the level of the corneal incision during cataract surgery. CDE will be recorded by the system.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Surgical, Study Director — Alcon Research, LLC
Locations (5):
- United States (5):
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Vance Thompson Vision, Sioux Falls, South Dakota
  - Whitsett Vision Group, Spring, Texas
  - Berkeley Eye Center, Sugar Land, Texas
  - The Eye Institute of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No